CLINICAL TRIAL: NCT00728897
Title: An Open Label, Randomised, Single Dose, Three-way Crossover Study to Investigate the Relative Bioavailability of a 100mg Capsule Compared to Four 25mg GSK598809 Capsules and the Effect of Food on the Pharmacokinetics of the 100mg Capsule in Healthy Male and Female Volunteers.
Brief Title: A Healthy Volunteer Study to Investigate the Relative Bioavailability of Two Forms of GSK598809 Capsules.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DAN111283
Record Dates: First submitted 2008-08-04; First posted 2008-08-06 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Substance Dependence
Keywords: Healthy volunteer; relative bioavailability.
MeSH Terms: conditions — Substance-Related Disorders

ARMS (6):
- Subjects receiving treatment sequence ABC (Experimental): Eligible subjects will receive treatment sequence ABC; A= 4x25 milligrams GSK598809 capsule given in fasted state, B= 100 milligrams GSK598809 capsule in given fasted state and C= 100 milligrams GSK598809 capsule given in fed state. The treatment sequence will be followed by at least a 7-day wash-out period between each dose.
  Interventions: Drug: GSK598809 new formulation; Drug: GSK598809 old formulation
- Subjects receiving treatment sequence ACB (Experimental): Eligible subjects will receive treatment sequence ACB; A= 4x25 milligrams GSK598809 capsule given in fasted state, C= 100 milligrams GSK598809 capsule given in fed state and B= 100 milligrams GSK598809 capsule in given fasted state. The treatment sequence will be followed by at least a 7-day wash-out period between each dose.
  Interventions: Drug: GSK598809 new formulation; Drug: GSK598809 old formulation
- Subjects receiving treatment sequence BAC (Experimental): Eligible subjects will receive treatment sequence BAC; B= 100 milligrams GSK598809 capsule in given fasted state, A= 4x25 milligrams GSK598809 capsule given in fasted state and C= 100 milligrams GSK598809 capsule given in fed state. The treatment sequence will be followed by at least a 7-day wash-out period between each dose.
  Interventions: Drug: GSK598809 new formulation; Drug: GSK598809 old formulation
- Subjects receiving treatment sequence BCA (Experimental): Eligible subjects will receive treatment sequence BCA; B= 100 milligrams GSK598809 capsule in given fasted state, C= 100 milligrams GSK598809 capsule given in fed state and A= 4x25 milligrams GSK598809 capsule given in fasted state. The treatment sequence will be followed by at least a 7-day wash-out period between each dose.
  Interventions: Drug: GSK598809 new formulation; Drug: GSK598809 old formulation
- Subjects receiving treatment sequence CAB (Experimental): Eligible subjects will receive treatment sequence CAB; C= 100 milligrams GSK598809 capsule given in fed state, A= 4x25 milligrams GSK598809 capsule given in fasted state and B= 100 milligrams GSK598809 capsule in given fasted state. The treatment sequence will be followed by at least a 7-day wash-out period between each dose.
  Interventions: Drug: GSK598809 new formulation; Drug: GSK598809 old formulation
- Subjects receiving treatment sequence CBA (Experimental): Eligible subjects will receive treatment sequence CBA; C= 100 milligrams GSK598809 capsule given in fed state, B= 100 milligrams GSK598809 capsule in given fasted state and A= 4x25 milligrams GSK598809 capsule given in fasted state. The treatment sequence will be followed by at least a 7-day wash-out period between each dose.
  Interventions: Drug: GSK598809 new formulation; Drug: GSK598809 old formulation

INTERVENTIONS:
Drug: GSK598809 new formulation — GSK598809 new formulation will be available as an immediate release capsule with a single dose of 100 milligrams, administered orally with 240 milliliters of water.
Drug: GSK598809 old formulation — GSK598809 old formulation will be available as an immediate release capsule with a single dose of 25 milligrams, administered orally with 240 milliliters of water.

SUMMARY:
Study to compare PK of a new 100mg capsule with four 25mg capsules. This is required because we plan to have only single capsules administered in the later phase clinical trials but we have not had a 100mg strength before. As this is a new previously untested strength we need to ensure that the PK is similar to that achieved using 4 x 25mg. The study will also assess the effect of high fat food on the PK of the 100mg capsule. The study is planned to consist of a single part , with three dosing periods, periods 1-3 consisting of 16 subjects. There will be a week wash out between each dose. In the three dosing periods subjects will either received 4x25 mg GSK598809 capsule in a fasted state, 100mg capsule in a fasted state or 100mg GSK598809 capsule in a fed state. Subjects will return to the centre for follow-up 7-14 days after the final dose. It is expected that the total duration of the study should be approximately eight weeks.

ELIGIBILITY:
Inclusion:

* Healthy as determined by responsible physician.
* Male or female between 18 to 65 years old.
* Females of non-child bearing potential and females of child-bearing potential that agree to use appropriate method of contraception for appropriate amount of time.
* Males that agree to use appropriate method of contraception for appropriate amount of time.
* Neither too fat nor too thin.
* Capable of giving written informed consent and being compliant with requirements within the informed consent.

Exclusion:

* Any current medical or psychiatric illness.
* Any history of chronic medical or psychiatric illnesses.
* Previous or current alcohol or drug abuse/dependence including nicotine.
* Female subjects must not be breastfeeding or been breastfeeding for a month.
* Serum prolactin exceeding normal range.
* Personal or family history of prolonged QTc syndrome.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-07-02 (Actual); Primary Completion 2008-07-29 (Actual); Study Completion 2008-07-29 (Actual)

PRIMARY OUTCOMES:
Blood sampling over a period of 96hrs post GSK598809 dosing in the three dosing periods. | Pre-dose, 0, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8. 10, 12, 16, 24, 48. 72 and 96 hours

SECONDARY OUTCOMES:
Safety and Tolerability: cardiovascular variables, vital signs, clinical labs, movement scales, prolactin, GH and TSH levels over 96 hours post dosing. Continuous adverse event monitoring from dosing until study conclusions. | Up to 96 hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

REFERENCES:
- See also: Results for study DAN111283 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/DAN111283?search=study&study_ids=DAN111283#rs